CLINICAL TRIAL: NCT06833632
Title: Detection of Circulating Tumour Cells, Spread Through Air Space and Lymph-nodal Micrometastasis in Patients With Lung Cancer Undergoing Surgical Resection With Curative Intent
Brief Title: Detection of Circulating Tumour Cells, Spread Through Air Space in Patients With Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: CTC22
Record Dates: First submitted 2024-11-28; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-10

CONDITIONS: Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Tissue samples will be evaluated for major NSCLC driver mutations by multigenic panels with NGS (next generation sequencing) and immunohistochemical expression of PDL1 will be tested on both primary tumour and CTC (only on the preoperative sample).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the prognostic impact of the presence of circulating tumour cells Circulating Tumour Cells (CTCs), Spread Through Air Space (STAS) and lymph node micrometastases in patients undergoing radical surgery for non-small cell lung neoplasia

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) is one of the leading causes of cancer deaths worldwide. Patients diagnosed with early-stage NSCLC are candidates for radical surgical resection with curative intent. However, disease recurrence after surgery is common, with 5-year recurrence rates ranging from about 20% in patients with stage I disease to about 50% in those with stage III disease. In detail, in patients operated with radical resection (R0), the loco-regional recurrence rate varies from 4.6 to 24%, with a significantly higher incidence in the first two years after surgery.

To date, only a few risk factors have been correlated with an increased propensity to develop recurrences, namely stage and some loco regional aggressiveness (e.g. pleural invasion, high-grade growth pattern, lymphovascular invasion), but there are still no certain elements that allow us to understand in advance the biology of the early spread of the disease and thus identify patients at high risk of relapse.

of relapse; the presence of these elements would have the potential advantage of playing a role both in recommending new therapeutic approaches for adjuvant treatment and in acting as biomarkers to anticipate the diagnosis or recurrence of lung cancer.

Until 2022, lobectomy was considered the standard of care for any type of lung neoplasm that was a candidate for surgery. Recent studies, however, have shown that even sublobar resections may allow adequate oncological radicality for tumours peripheral tumours of small size (<2 cm) . Moreover, in the last decade, technological development has allowed a gradual replacement of traditional open techniques with mini-invasive techniques (videothoracoscopy, Video Assisted Thoracic Surgery (VATS), or robotic, Robotic Assisted Thoracic Surgery (RATS)).

Circulating tumour cells (CTCs) are considered to be the site of origin for possible disease recurrence in several cancers, showing a higher rate of disease recurrence in the case of high CTC levels. Despite this, their specific clinical role in lung cancer has not yet been clarified. CTCs from the peripheral blood of patients with breast cancer, melanoma, NSCLC and small cell lung cancer can form tumours in mice immunocompromised mice, confirming their carcinogenic potential. Furthermore, the presence of CTCs has also been correlated with manipulation of the lung during surgery, which would seem to favour dissemination, although the clinical significance is uncertain.

Recent studies have highlighted the importance of the molecular profile of neoplasms lung neoplasms that could change the standard of care with regard to neoadjuvant or adjuvant therapies. Molecular assessment is usually performed on biopsies or on the operative specimen of the primary tumour, but could potentially be performed on circulating tumour cells. Weak evidence on the clinical role of CTCs also includes their role in defining the molecular profile of the tumour.

In addition to haematogenous spread of which CTCs could be a warning sign, NSCLC can potentially spread via the airway and lymphatic route. Spread via the airway and through the alveolar spaces has recently been observed, especially in the adenocarcinoma histotype, and codified by the World Health Organisation (WHO 2021) as Spread Through Air Space (STAS); as for lymphatic invasion lymphatic invasion, in addition to intrapulmonary lymphatic vessel invasion, it is manifested by the presence of lymph node metastases or micrometastases.

In detail, STAS are defined as tumour cells existing within alveolar spaces in the lung parenchyma beyond the edge of the main neoplasm, in close proximity to the edge of the main neoplasm. STAS can be found mainly, but not only, in lung adenocarcinomas and in about 35-40% of early stage clinical NSCLC; some studies have shown their correlation with a worse prognosis than in patients without STAS .

Micrometastases, in other body districts such as breast and axillary locoregional lymph node metastases, on the other hand, are defined as tumour aggregates between between 0.2 and 2.0 mm. In the literature, data on the incidence of lymph node micrometastases in NSCLC are inconsistent and range from 10-80%. Compared to patients with macroscopic lymph node involvement, micrometastases seem to be related to a better prognosis, but, on the other hand, outcomes seem to be worse than in N0 pathological patients.

The objectives of the study are to :

1. Check whether the presence and/or levels of CTC is associated with disease-free survival (DFI)
2. To assess the pattern of recurrence in patients with CTC, STAS and lymph node micrometastases

Secondary objectives

1. Quantify the difference in intraoperative release of CTC into the bloodstream based on the intraoperative variables:

   * Resection sequence of the hilar structure (first vein or artery)
   * Lung management according to different surgical techniques (open, VATS, RATS)
   * Type of resection: segmentectomy, lobectomy, pneumonectomy
2. Check for association between CTC, presence of STAS and presence of lymph node micrometastases
3. Check whether the presence and/or levels of CTC, STAS and lymph node micrometastases are associated with long-term outcomes (DFI, OS)
4. Compare the molecular profile of CTCs and the primary tumour

ELIGIBILITY:
Inclusion Criteria:

* obtaining voluntary written informed consent
* diagnosis of NSCLC
* clinical stage I-IIA cN0
* Candidates for surgical resection

Exclusion Criteria:

* Pregnancy
* Induction therapy for pulmonary neoplasia
* Patients who have received systemic treatment for previous cancers in the last three years prior to lung surgery
* Any previous surgery for lung cancer
* Patients with other active neoplasms
* Infiltration of the chest wall

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is low-risk, human-tissue, prospective, single-center experimental study conducted on patients undergoing surgery for removal of stage I-IIA NSCLC.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2025-09-11 (Estimated); Study Completion 2025-09-11 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Through study completion, up to 36 months.
  Overall survival (in months) will be assessed for each patient enrolled in the study from the day of surgery to the last follow-up or death whichever comes first
Disease-free survival (DFS) | Through study completion, up to 36 months.
  DFS (in months) will be assessed for each patient enrolled in the study: the relapse is defined as the first evidence of recurrence of disease on instrumental examinations instrumental examinations performed in the follow-up.
Global recurrence rate | Through study completion, up to 36 months.
  Percentage of patients with any recurrence
Type of recurrence | Through study completion, up to 36 months.
  Number of patients with local, regional distant or multiple recurrence

SECONDARY OUTCOMES:
Circulating Tumour Cells (CTC) | Through study completion, the day before surgery and 30 days after surgery, up to 36 months.
  Presence or absence, level of CTCs measured as median value with interquartile range
Spread through air space (STAS) | Through study completion, at the time of pathological analysis of surgical specimen (approximately 36 months)
  Presence or absence of STAS
Micrometastases at lymph nodes | Through study completion, at the time of pathological analysis of surgical specimen (approximately 36 months)
  Presence or absence of micrometastasis
Molecular mutations in EGFR, ALK, ROS1, KRAS genes | Through study completion, at the time of pathological analysis of surgical specimen (approximately 36 months)
  Counting of mutations though multigenic panels
PD-L1 expression | Through study completion, at the time of pathological analysis of surgical specimen (approximately 36 months)
  Assessment of level of expression of PD-KL1 gene in CTCs and tumour

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Bertoglio, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS - Azienda Ospedaliero Universitaria di Bologna, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: Undecided